CLINICAL TRIAL: NCT02222025
Title: Injury Prevention in Children´s Football (FIFA 11+ Kids): a Cluster-randomized Controlled Trial
Brief Title: Injury Prevention in Children´s Football
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Basel (Other)
Collaborators: VU University of Amsterdam (Other); Charles University, Czech Republic (Other); Universität des Saarlandes (Other); FIFA-Medical Assessment and Research Centre (F-MARC) (Unknown)
Responsible Party: Principal Investigator, Oliver Faude, Dr., University of Basel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2014-232
Record Dates: First submitted 2014-08-14; First posted 2014-08-21 (Estimated); Last update posted 2016-04-22 (Estimated); Status verified 2016-04

CONDITIONS: Football Injuries in Children

ARMS (2):
- Injury Prevention Programme (Experimental): see intervention prescription
  Interventions: Other: Injury Prevention Programme
- Control (No Intervention): The coaches of the control group will receive the instruction to regularly perform a common warm-up consisting of running and ball-based exercises (sham treatment, no neuromuscular and stability exercises).

INTERVENTIONS:
Other: Injury Prevention Programme — The injury prevention program will be included at the beginning of the usual football training by replacing the traditional warm-up. The programme will be conducted by the coaches at least two times a week (with exception of school holidays). The prevention programme contains seven exercises and lasts about 15 min after familiarisation. Three exercises focus on unilateral, dynamic stability of the lower extremities (hopping, jumping and landing). Further, three exercises emphasize whole body and trunk stability. The last exercise contains rolling movements to improve fall technique. The difficulty of each exercise can be progressively increased in five steps. Players start at the level of difficulty which corresponds to their current performance level. They will proceed to the next level when they perform the exercises with good control. This will be assessed by the coaches.
  Arms: Injury Prevention Programme

SUMMARY:
Playing football can induce considerable beneficial health effects, but is also a high-intensity and high-impact sport with many situations of direct contact between players which bear the risk of injury. Thus, it is necessary to implement preventive measures to reduce the risk of injury and support the health benefits.

Injury characteristics of players older than 13 years are similar to adult players and, thus, similar preventive measures are beneficial. Younger players seem to show partly different injury characteristics. Consequently, preventive programmes proven effective in late adolescent or adult players need to be adapted for younger age groups. To date, no study investigated the prevention of football injuries in children under the age of 13 years.

We aim to assess the effectiveness of an exercise-based prevention program to reduce football-related injuries in children younger than 13 years.

The primary outcome in this study is the overall injury rate. Secondary outcomes are the rate of severe injuries and acute injuries.

The study is designed as a two-armed cluster-randomized controlled trial. We will recruit 9 to 12 years old children (boys and girls, born 2002 to 2005) participating in regular training and match play in an officially registered football club in Switzerland (further study centres are located in the Netherlands, Germany and the Czech Republic). The chosen age group is usually subdivided into two age categories (9/10 years, 11/12 years).

Recruitment will take place via the national and regional football associations.

Inclusion criteria are: the clubs must be officially registered in the regional football association, children must be between 9 and 12 years old at the start of the study and regular training must take place at least twice per week. Teams will be excluded, if the coaches already perform a structured warm-up focusing on neuromuscular control or an existing injury prevention programme.

Injury surveillance will include a baseline questionnaire, players´ exposure and injury registration. Anthropometric baseline data and information regarding previous football-related injuries will be obtained prior to the start of the study from the parents. Injury and exposure surveillance will be assisted by an automated internet-based injury recording system which has been developed and applied during our own epidemiological project.

For all participating teams, one contact person will be appointed. Those persons will be provided with exact instructions on injury definitions as well as examples how to complete the injury and exposure forms within the online injury recording system.

If an injury occurred, one trained person will contact the coach as well as the player and the parents by telephone and/or e-mail to assess all relevant aspects of the injury based on a standardized injury registration form. In case of injuries which require medical treatment parents will be supported to receive the exact diagnosis from the attending physician (either as specific written diagnosis or by use of a specific injury coding system). Two blinded investigators will additionally assess all information with regard to each injury to allow for objective and independent injury surveillance.

20 study assistants and 4 scientific assistants will support coaches with data collection and injury recording. Each study assistant will be responsible for eight clubs. Study assistant will regularly keep in touch with the clubs and will visit two training sessions of each team during the study period.

The intervention period will last one complete season. The injury prevention program will be included at the beginning of the usual football training by replacing the traditional warm-up. The programme will be conducted at least two times a week by the intervention teams. The prevention programme contains seven exercises and lasts about 10 to 15 min after familiarisation. Three exercises focus on unilateral, dynamic stability of the lower extremities (hopping, jumping and landing). Further, three exercises emphasize whole body and trunk stability. The last exercise contains rolling movements to improve fall technique.

The coaches of the control group will receive the instruction to regularly perform a common warm-up consisting of running and ball-based exercises (sham treatment, no neuromuscular and stability exercises).

The yearly incidence injured players in children is 8.6%. A risk reduction of one third has been recently acknowledged as a relevant effect size for injury rate. This corresponds to a reduction of the yearly incidence to 5.8% injured players. In order to achieve a statistical power of 80% and taking an allocation ratio of 1:1 and a cluster-inflation factor of 1.7 into account, in total 4´000 players are needed for statistical analysis. Assuming a realistic drop-out rate of about 33%, 6´000 children will be initially recruited.

ELIGIBILITY:
Inclusion Criteria:

* officially registered football club in the regional football association,
* children must be between 9 and 12 years old at the start of the study
* regular training must take place at least twice per week

Exclusion Criteria:

* a structured warm-up focusing on neuromuscular control or an existing injury prevention programme is already performed

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3895 (Actual)
Dates: Start 2014-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Overall injury rate | up to 12 months

SECONDARY OUTCOMES:
Rate of severe injuries and acute injuries | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Sport, Exercise and Health, University of Basel, Basel, Switzerland

REFERENCES:
- [Derived] Beaudouin F, Rossler R, Aus der Funten K, Bizzini M, Chomiak J, Verhagen E, Junge A, Dvorak J, Lichtenstein E, Meyer T, Faude O. Effects of the '11+ Kids' injury prevention programme on severe injuries in children's football: a secondary analysis of data from a multicentre cluster-randomised controlled trial. Br J Sports Med. 2019 Nov;53(22):1418-1423. doi: 10.1136/bjsports-2018-099062. Epub 2018 Oct 2. PMID 30279219
- [Derived] Rossler R, Junge A, Bizzini M, Verhagen E, Chomiak J, Aus der Funten K, Meyer T, Dvorak J, Lichtenstein E, Beaudouin F, Faude O. A Multinational Cluster Randomised Controlled Trial to Assess the Efficacy of '11+ Kids': A Warm-Up Programme to Prevent Injuries in Children's Football. Sports Med. 2018 Jun;48(6):1493-1504. doi: 10.1007/s40279-017-0834-8. PMID 29273936